CLINICAL TRIAL: NCT06304974
Title: A Phase Ill Randomized Controlled Clinical Study Comparing BL-B01D1 With Chemotherapy of Physician's Choice as Second Line Treatment in Patients With Recurrent or Metastatic Esophageal Squamous Cell Carcinoma After Failure of PD-1/PD-L1 Monoclonal Antibody in Combination With Platinum-based Chemotherapy
Brief Title: A Study Comparing BL-B01D1 With Chemotherapy of Physician's Choice in Patients With Recurrent or Metastatic Esophageal Squamous Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BL-B01D1-305
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Irinotecan; Paclitaxel; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Participants receive BL-B01D1 as intravenous infusion for the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: BL-B01D1
- Control group (Experimental): Participants receive Irinotecan or paclitaxel or docetaxel in the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: Irinotecan; Drug: paclitaxel; Drug: docetaxel

INTERVENTIONS:
Drug: BL-B01D1 — Administration by intravenous infusion
  Other Names: iza-bren; izalontamab brengitecan; BMS-986507
  Arms: Experimental Group
Drug: Irinotecan — Administration by intravenous infusion
  Arms: Control group
Drug: paclitaxel — Administration by intravenous infusion
  Arms: Control group
Drug: docetaxel — Administration by intravenous infusion
  Arms: Control group

SUMMARY:
This study is a registered phase Ill, randomized, open-label, multicenter study to evaluate the efficacy and safety of BL-B01D1 in patients with recurrent or metastatic esophageal squamous cell carcinoma after failure of PD-1/PD-L1 monoclonal antibody in combination with platinum-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent and follow the requirements of the protocol;
2. Age ≥18 years old;
3. Expected survival time ≥3 months;
4. Patients with recurrent or metastatic esophageal squamous cell carcinoma confirmed by histology or cytology;
5. Consent to provide archival tumor tissue samples or fresh tissue samples of primary or metastatic lesions within 3 years;
6. Must have at least one measurable lesion according to RECIST v1.1 definition;
7. ECOG 0 or 1;
8. Toxicity of previous antineoplastic therapy has returned to ≤ grade 1 defined by NCI-CTCAE v5.0;
9. No severe cardiac dysfunction, left ventricular ejection fraction ≥50%;
10. No blood transfusion and no use of any cell growth factor drugs were allowed within 14 days before randomization, and the level of organ function had to be adequate;
11. Urine protein ≤2+ or < 1000mg/24h;
12. A serum pregnancy test must be performed within 7 days before the start of treatment for premenopausal women who are likely to have children, and the result must be negative and must not be lactating; All enrolled patients should take adequate barrier contraception during the entire treatment cycle and for 6 months after the end of treatment.

Exclusion Criteria:

1. Chemotherapy, targeted therapy, biological therapy, etc., had been used within 4 weeks or 5 half-lives before randomization, and palliative radiotherapy and modern traditional Chinese medicine preparations approved by NMPA had been used within 2 weeks;
2. Patients with recurrent esophageal squamous cell carcinoma suitable for radical local treatment should be excluded;
3. Frontline received ADCs with topoisomerase I inhibitors as toxins;
4. History of severe heart disease and cerebrovascular disease;
5. Prolonged QT interval, complete left bundle branch block, III degree atrioventricular block, frequent and uncontrollable arrhythmia;
6. diagnosed with active malignancy within 3 years before randomization;
7. Hypertension poorly controlled by two antihypertensive drugs;
8. patients with poor glycemic control;
9. present with grade ≥1 radiation pneumonitis according to the RTOG/EORTC definition; A previous history of interstitial lung disease (ILD) or a suspicion of such disease on imaging during screening;
10. Complicated with pulmonary diseases leading to clinically severe respiratory function impairment;
11. patients with active central nervous system metastases;
12. Severe infections within 4 weeks before randomization; Evidence of pulmonary infection or active pulmonary inflammation within 2 weeks before randomization;
13. patients with massive or symptomatic effusions or poorly controlled effusions;
14. Imaging examination showed that the tumor had invaded or wrapped around the large blood vessels in the abdomen, chest, neck, and pharynx;
15. serious unhealed wounds, ulcers, or fractures, or clinically significant bleeding or obvious bleeding tendency within 4 weeks before signing the informed consent;
16. patients with inflammatory bowel disease, extensive bowel resection history, immune enteritis history, intestinal obstruction or chronic diarrhea;
17. patients with a history of allergy to recombinant humanized antibodies or to any of the excipients of BL-B01D1;
18. had a history of autologous or allogeneic stem cell transplantation;
19. Human immunodeficiency virus antibody positive, active hepatitis B virus infection or hepatitis C virus infection;
20. a history of severe neurological or psychiatric illness;
21. received other unmarketed investigational drugs or treatments within 4 weeks before randomization;
22. subjects scheduled for vaccination or who received live vaccine within 28 days before study randomization;
23. Other circumstances in which the investigator considered it inappropriate to participate in the trial because of complications or other circumstances.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 497 (Actual)
Dates: Start 2024-03-19 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 24 months
  Progression-free survival (PFS) as assessed by BIRC is defined as the time between the date subjects are randomized and the first observation of disease progression (based on BICR's image-based assessment) or death.
Overall survival (OS) | Up to approximately 24 months
  Overall survival (OS) is defined as the time between the subject's randomization date and subject's death.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 24 months
  Objective response rate (ORR) is defined as the number of CR and PR in the treatment and control groups divided by the number of that group in the full analysis set (FAS).
Disease Control Rate (DCR) | Up to approximately 24 months
  Disease Control Rate (DCR) : Percentage of all randomized subjects who rated the best overall response (BOR) as complete response (CR), partial response (PR), and disease stabilization (SD) according to RECIST 1.1 criteria.
Duration of Response (DOR) | Up to approximately 24 months
  Duration of Response (DOR) : defined as the period from the date when tumor response is first recorded to the date when objective tumor progression is first recorded or the date of death.
Treatment Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of BL-B01D1. The type, frequency and severity of TEAE will be evaluated during the treatment of BL-B01D1.
Cmax | Up to approximately 24 months
  Maximum serum concentration (Cmax) of BL-B01D1 will be investigated.
T1/2 | Up to approximately 24 months
  Half-life (T1/2) of BL-B01D1 will be investigated.
Anti-drug antibody (ADA) | Up to approximately 24 months
  Frequency of anti-BL-B01D1 antibody (ADA) will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, PHD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China